CLINICAL TRIAL: NCT06617481
Title: RhPSMA-7.3(18F)-PET Scan to Detect Prostate Cancer in Patients with Early PSA Recurrence
Brief Title: PET Scan Study to Detect Prostate Cancer in Patients with Early PSA Recurrence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AdventH; IRBNet # 2067493 (Other: AdventHealth)
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer (Post Prostatectomy)
Keywords: Rising PSA following cancer prostatectomy surgery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Main Arm (Other): Single Arm receiving PET scan with 18F-rhPSMA-7.3 (Posluma)
  Interventions: Drug: 18F-rhPSMA-7.3 (Posluma)

INTERVENTIONS:
Drug: 18F-rhPSMA-7.3 (Posluma) — PET Scan using Posluma for detection of early recurrence of prostate cancer.

SUMMARY:
Flotufolastat F-18, sold under the brand name Posluma, is a radioactive diagnostic agent for use with positron emission tomography (PET) imaging for prostate cancer.

The research is being done to study the capability of 18F-rhPSMA-7.3 (flotufolastat F-18) PET scan to detect prostate cancer when there are very low levels of Prostate-Specific Antigen (PSA) following previous radical prostatectomy surgery.

DETAILED DESCRIPTION:
This is not an investigational study drug. Flotufolastat PET scan is FDA Approved for positron emission tomography (PET) of prostate-specific membrane antigen (PSMA) positive lesions in men with prostate cancer with suspected metastasis who are candidates for initial definitive therapy and those with suspected recurrence based on elevated serum prostate-specific antigen (PSA) level. In this research study, the flotufolastat-PET scan will be repeated if the initial scan does not show cancer and if PSA further rises by greater than 0.1 ng/ml. Other currently used scans for this purpose do not detect cancer in all patients with low levels of rising PSA.

ELIGIBILITY:
Inclusion Criteria:

* History of localized adenocarcinoma of the prostate with prior curative intent radical prostatectomy.
* An elevated PSA test result that is greater than or equal to 0.1 ng/ml and less than 0.5

Exclusion Criteria:

* Patients who are planned to have an x-ray contrast agent or other PET radiotracer & less than 24 hours prior to the flotufolastat F-18 PSMA-PET scan.
* Patients currently receiving Androgen Deprivation Therapy (ADT).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-09-05 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate | 24 months
  Patients who undergo at least one rhPSMA-7.3 (18F) PET-scan will be analyzed for the primary endpoint. The malignant lesion detectability rate will be summarized using percentage and 95% confidence interval estimates overall and for those who underwent a single scan or both scans. The diagnostic evaluation aims to identify individuals who are most likely to have an isolated local relapse, as they have the most significant potential for achieving long-term disease control through additional local therapy.

SECONDARY OUTCOMES:
Correlation with biopsy | 24 months
  In those patients who undergo biopsy of a lesion, correlation with pathology report diagnosis will be reviewed.
Correlation with other imaging modalities | 24 months
  In those patients who undergo other imaging modalities to confirm the results of the rhPSMA-7.3 (18F) PET-scan, correlation with other imaging modalities will be reviewed.
Response to therapy | 24 months
  In those patients who undergo cancer directed therapy with radiation alone or with androgen deprivation therapy, the follow-up PSA test values after therapy will be reported.
Adverse Events | 24 hours
  Safety and toxicity data will be collected to evaluate any patient reported adverse effects. Safety Follow-up Call Within 24 hours of each Injection/Scan

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Decision to be made at the end of enrollment period of 30 patients